CLINICAL TRIAL: NCT04255251
Title: Effectiveness Silver Diamine Fluoride Versus Sodium Fluoride in Arresting Caries Around Crown Margins in Older Adults
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of New England (Other)
Responsible Party: Principal Investigator, Shaista Rashid, Assistant Clinical Professor, University of New England
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Universityof New Engalnd
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Caries Roots; Flouride Varnish; Caries; Dentin; Caries Arrested
MeSH Terms: conditions — Root Caries | interventions — silver diamine fluoride; Fluorides, Topical

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly into treatment and control group using a predetermined randomization protocol.
Who Masked: Participant, Investigator
Masking Description: Participants will not know which type of fluoride they are getting around their crow margins.
  Principal investigator will measuring the extend of the decay does not know about the type of fluoride treatment patient got.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Subjects in this group will receive Silver Diamine Fluoride around their crown margins every six month for the next 3 years.
  Interventions: Drug: Silver Diammine Fluoride
- Fluoride varnish group (Active Comparator): Subjects in this group will receive fluoride varnish around their crown margins every six month for the next 3 years.
  Interventions: Drug: Fluoride Varnishes

INTERVENTIONS:
Drug: Silver Diammine Fluoride — Subjects will receive SDF around their crown margins every 6 months for next 3 years.
  Arms: Intervention group
Drug: Fluoride Varnishes — Subjects will receive SDF around their crown margins every 6 months for next 3 years.
  Arms: Fluoride varnish group

SUMMARY:
Dental caries is a multifactorial, progressive disease which is the major causes of dental pain, infection and tooth loss. Dental caries can substantially compromise the quality of life in older adults 1 2. As the number of older adults in the US increases, the dental professionals have become increasingly concerned with the dental need of elderly and preventive regimes to reduce the incidence of caries3 .

Prevention becomes an area of paramount importance. Many studies have advocated nonsurgical intervention for shallow dentin caries lesion.The most effective method for prevention to date is considered to be fluoride. In the United states fluoride has been incorporated in many ways like water fluoridation, fluoride mouth wash, dentifrices and professionally applied fluoride varnishes . The American Dental Association (ADA) recommended the use of fluoride for patients of all ages who are at risk of developing dental caries7 . With the high success of fluoride, another treatment method using Silver Diamine Fluoride (SDF) is gaining popularity in the United States. SDF has been used in many countries like Japan, Australia, China, and Cuba for treatment of caries . Successful treatment data from other countries is promising, and promoting the use of SDF in the United States. SDF is available in the United States as 38% aqueous solution and approved as a desensitizing agent. American Dental Association published an evidence-based clinical practice guideline on nonrestorative treatments for caries teeth and recommended use of SDF on a carious cavitated lesion on permanent teeth9 . Clinical studies have shown the effectiveness of SDF in arresting root caries in older adults.

DETAILED DESCRIPTION:
Potential subjects will be identified through regular appointments. Screening will be performed on subjects to determine their eligibility based on inclusion and exclusion criteria. Subjects will sign an informed consent before enrollment in the study. Patient will be receiving one of the two fluoride treatments, Silver Diamine Fluoride or Sodium fluoride, to arrest caries around crown margins. Clinical and radiographic exam will be performed on all the participants.

Clinical exam will include the following

1. DIAGOdent:
2. Tectile exam:

The procedures of every clinical appointments will be as following:

First appointment:

Visit will include

* Health history
* Caries risk assessment
* Clinical exam (DIAGNOdent, tactile) (described above)
* Radiograph (described above)
* Subject will sigh consent form
* Treatment group will receive SDF
* Control group will receive Fluoride varnish

Second visit (6 month from the first appointment ):

Visit will include

* Health history retake
* Caries risk assessment retake
* New Clinical exam (DIAGNOdent, tactile)
* New Radiograph
* Subject will receive his or her treatment according to their allocation

Third visit (12 month from the first appointment ):

Visit will include

* Health history retake
* Caries risk assessment retake
* New Clinical exam (DIAGNOdent, tactile)
* New Radiograph
* Subject will receive his or her treatment according to their allocation

Third visit (12 month from the first appointment ):

Visit will include

* Health history retake
* Caries risk assessment retake
* New Clinical exam (DIAGNOdent, tactile)
* New Radiograph
* Subject will receive his or her treatment according to their allocation

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years old with crown/bridges
* Open crown margins
* Decay present around crown margins
* Pt is not intention to go with the conventiontial restorative treatment to replace the crown for any reason
* Subjects who can do the follow up for at least one year

Exclusion Criteria:

* Teeth with periapical lesion
* Teeth which have pain to percussion
* Subjects who have silver or fluoride allergy
* Subjects who have gingivitis
* Subjects who have stomatitis
* Subjects who have tooth mobility
* Subjects who have furcation involvement

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Tactile exam to evaluate extend of caries around tooth margin | Every 6 month for next 3 years
  WHO ball end probe will be used to detect cavities around the restoration margins.
  Code 0: Sound tooth surface with restoration Code 1: First visual change in enamel Code 2: Distinct visual change in enamel/ dentin adjacent to restoration Code 3: Carious defect of more than 0.5 mm Code 4: Marginal caries in enamel/dentin/cementum adjacent to restoration with dark shadow Code 5: Distinct cavity adjacent to restoration Code 6: Extensive distinct cavity with visible dentine

SECONDARY OUTCOMES:
DIAGOdent: laser fluorescence to aid in the detection of caries | Every 6 month for next 3 years
  As the incident laser light is dispersed into the site, carious tooth structure will exhibit fluorescence, proportionate to the degree of caries, resulting in elevated scale readings on the display. Healthy tooth structure exhibits little or no fluorescence and will result in very low scale readings on the display. Over 90% accurate in detecting lesions not detectable with an explorer or bitewing X-rays. The remote display for DIAGNOdent pen uses infra-red signals, and the values are shown simultaneously on the DIAGNOdent pen and on the remote display

CONTACTS AND LOCATIONS:
Locations (1):
- University of New England, Portland, Maine, United States

REFERENCES:
- [Background] Giusti L, Steinborn C, Steinborn M. Use of silver diamine fluoride for the maintenance of dental prostheses in a high caries-risk patient: A medical management approach. J Prosthet Dent. 2018 May;119(5):713-716. doi: 10.1016/j.prosdent.2017.06.007. Epub 2017 Sep 6. PMID 28888414
- [Result] Seifo N, Cassie H, Radford JR, Innes NPT. Silver diamine fluoride for managing carious lesions: an umbrella review. BMC Oral Health. 2019 Jul 12;19(1):145. doi: 10.1186/s12903-019-0830-5. PMID 31299955